CLINICAL TRIAL: NCT03211091
Title: Prove/Cerebrovascular Registry
Brief Title: Cerebrovascular Registry
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mohammad Saadatnia, Professor Mohammad Saadatnia, Isfahan University of Medical Sciences
Other Study IDs: Prove registry
Record Dates: First submitted 2017-04-24; First posted 2017-07-07 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Cerebrovascular Disorders
MeSH Terms: conditions — Cerebrovascular Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with stroke were registered based on the WHO/ MONICA protocol and were followed-up for 28 days, starting in 2015 in PROVE Registry

DETAILED DESCRIPTION:
PROVE program started in 2015, the registration of stroke continued but followed the WHO Stepwise method instead of WHO/MONICA .Patients are followed up for two years. The corresponding questionnaire covered the patients' demographic data, medical history upon hospital admission, history of comorbidities, medications used prior to the treatment, history of drug abuse, heart and brain imaging, history of blood tests and blood diseases, hospital treatments received, hospitalization complications, medications prescribed at the time of discharge, discharge status and the definite diagnosis of type of stroke according to CT or MRI.

The patients were followed-up over the phone or in person from the 1st, 3rd and 12th months to two years. The patients' disabilities were measured using the Barthel Index and the Modified Rankin Scale (MRS). The reliability and validity of these two questionnaires have already been investigated in Persian. In addition, secondary prevention measures, rehabilitation status and the incidence of new cardiovascular events were also examined in the follow-up. The stroke registration personnel received an initial training of three two-hour sessions and monthly one-hour retraining sessions. They visited the archives of various hospitals on a daily basis and registered the data contained in the records

ELIGIBILITY:
Inclusion Criteria:

* patients with acute Stroke (Hemorrhagic and Non Hemorrhagic)

Exclusion Criteria:

* patients who do not agree to continue cooperation
* patients with incomplete documents

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with stroke or stroke history
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-01-10 (Actual); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
disability | 3 months
  the Barthel Index

SECONDARY OUTCOMES:
rehabilitation | 3 months
  Ashworth Scale
rehabilitation | 12 months
  Modified Ashworth Scale

IPD SHARING:
Plan to Share IPD: Undecided